CLINICAL TRIAL: NCT02639260
Title: A Phase 1 Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ManNAc in Subjects With Primary Podocyte Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160036; 16-DK-0036
Record Dates: First submitted 2015-12-23; First posted 2015-12-24 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Kidney Disease
Keywords: Nephrotic Syndrome; Glomerular Filtration Rate; Sialic Acid; Proteinuria
MeSH Terms: conditions — Kidney Diseases; Nephrotic Syndrome; Proteinuria | interventions — N-acetylmannosamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): 3,000 mg/day
  Interventions: Drug: N-acetyl D-mannosamine
- Cohort B (Experimental): 10,000 mg/day
  Interventions: Drug: N-acetyl D-mannosamine

INTERVENTIONS:
Drug: N-acetyl D-mannosamine — dose escalation

SUMMARY:
Three kidney diseases that affect both children and adults are minimal change disease (MCD), focal segmental glomerulosclerosis (FSGS) and membranous nephropathy (MN). These diseases are characterized by proteinuria (protein in the urine) and in the cases of FSGS and membranous nephropathy, a tendency to progressive scarring of the glomerulus (the filtering units of the kidneys) that leads to end-stage kidney disease. Several therapies are available for these diseases, but these therapies do not provide lasting reduction in proteinuria for many subjects. In the current study, carried out at the NIH Clinical Center, we are testing a new therapy, ManNAc. ManNAc is a naturally occurring uncharged sugar that cells use to produce negatively charged sialic acid. Kidney cells attach sugars such as sialic acids to proteins and lipids (resulting in glycans), and these assist in cell function. Mouse models of the inherited muscle disease GNE myopathy, which is due to sialic acid deficiency on muscle glycans, responded favorably to oral ManNAc therapy and a clinical trial of ManNAc is ongoing in GNE myopathy subjects. There is evidence that some subjects with MCD, FSGS or MN do not put enough sialic acids on glomerular proteins and so ManNAc therapy may increase sialic acid production and sialylation of glomerular proteins in these subjects. For the present study, we will recruit 12 subjects who have MCD, FSGS or MN. Each subject will stay at the NIH Clinical Center for 11 days to receive oral ManNAc. The primary purposes of the study are to determine: 1) the safety of ManNAc in subject s with kidney disease; and 2) the ManNAc and sialic acid metabolism related to ManNAc in subjects with kidney disease. Concentrations of ManNAc and sialic acid will be measured in plasma at various times before and after dosing. If this study suggests that ManNAc is safe in subject with kidney disease, the results will be used to plan a longer-term study to determine whether it is effective at reducing proteinuria....

DETAILED DESCRIPTION:
Background. ManNAc (N-acetyl D-mannosamine) is an uncharged monosaccharide that is the biologic precursor of N-acetyl neuraminic acid (Neu5Ac, sialic acid). Sialic acids are the negatively charged, terminal monosaccharides of carbohydrate chains that are attached to glycoproteins and glycolipids (glycans). Most glycans serve cellular signaling functions, and frequently appear on the cell surface or are secreted into the circulation. ManNAc is currently in development as a therapy for the rare muscular dystrophy, GNE Myopathy (also called HIBM, hereditary inclusion body myopathy), caused by deficiency of GNE, the key enzyme in sialic acid synthesis (clinicaltrials.gov; NCT01634750).

A Phase 1a trial was completed and a Phase 2 trial for ManNAc for GNE myopathy subjects has been initiated through efforts of NCATS (TRND program; PI: Dr. Carrillo-Carrasco) and NHGRI (Dr. Huizing, Dr. Malicdan; Sponsor: Dr. Gahl), most of whom are Associate Investigators on this protocol. The NHGRI basic research group has documented podocytopathy, glomerular protein hyposialylation and severe proteinuria in mice deficient in GNE and found that their podocyte ultrastructure improved, sialylation increased and proteinuria decreased with oral ManNAc therapy. Human kidney biopsy tissue from subjects with various primary podocyte diseases, including minimal change disease (MCD), focal segmental glomerulosclerosis (FSGS) and membranous nephropathy (MN), also showed glomerular hyposialylation (manuscript in preparation).

Purpose. We propose to carry out a Phase 1 escalating dose study to evaluate the safety, tolerability, and pharmacokinetics of ManNAc in nephrotic subjects with primary podocyte diseases.

Subjects. We propose to enroll 12 subjects with MCD, FSGS or MN. Up to 24 total subjects may be enrolled to accomodate screening failures and withdrawals, for a total of 12 subjects receiving at least one dose of the study drug. We will recruit subjects in 4 groups (2-3 subjects each) grouped by estimated glomerular filtration rate (eGFR).

Intervention. This dose escalation study will involve two progressive ManNAc dose cohorts (each with N= 6) of 3,000 mg/day and 6,000 mg/day. Drug exposure will occur in a single dose phase, involving one dose of oral ManNAc followed by a 72 hour pharmacokinetics and safety study, and a multiple dose phase, involving ManNAc administered two times/day for 5 days. Dose escalation will occur when the lower dose is assessed safe in all subjects by a Safety Review Committee.

Outcomes. We will assess safety by self-reported symptoms and by standard laboratory testing. Pharmacokinetics will be analyzed using plasma ManNAc and Neu5Ac (sialic acid) levels. The effects of reduced eGFR on these parameters will be assessed. While the study duration is short and there is no placebo control, the effect of ManNAc therapy on proteinuria, from the baseline to the end of the extension phase, will be examined on a research basis.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Kidney biopsy manifesting MCD, FSGS (including collapsing glomerulopathy) or MN. Prior kidney biopsy is a requirement for inclusion. Kidney biopsy materials will be reviewed by NIH pathology (Dr. Avi Rosenberg, or another member of his team in his absence) to confirm the diagnosis. With regard to FSGS, all histologic variants, including collapsing, tip, cellular, perihilar and NOS will be included; primary, adaptive, and genetic FSGS will be included; viral-associated and drug-associated FSGS will be excluded. The rationale for including multiple primary nephrotic diseases is that the pharmacokinetics is likely to be similar and all these diseases have a need for effective therapy with low toxicity profile.
  2. Age >18 years weighing more than 40 kg of either sex. The rationale for excluding children is that we lack safety data for patients with nephrotic and/or reduced GFR and that we have no evidence for benefit in proteinuric subjects.
  3. Subjects must either not be taking immunosuppressive therapy (e.g., prednisone, cyclosporine, tacrolimus or mycophenolate mofetil) or, alternatively, be able to tolerate a stable dose of such a therapy from day -30 to day +31. If medically necessary, immunosuppressive therapy will be adjusted during the study. Subjects who are on renin angiotensin pathway inhibitor therapy will not be asked to discontinue their current regiment and will be included in the study.
  4. Weight >40 kg. Subjects 40-50 kg will only be placed in the low-dose Cohort A. Subjects >50 kg can be placed in either Cohort A (3,000 mg/day) or Cohort B (6,000 mg/day). The rationale is to adhere to the maximum allowable starting dose of 193.5 mg DEX-M74/kg body weight/day, derived from preclinical animal toxicology studies.
  5. Subjects with random void urine protein/creatinine ratio > 1 g/g.
  6. Subjects with an estimated glomerular filtration rate (eGFR) .15 mL/min/1.73 m^2 will be included. The rationale is that we wish to determine the effect of eGFR on ManNAc and Neu5Ac (sialic acid) metabolism (including plasma PK). We will compare 2 eGFR groups: subjects with stage 4 CKD (eGFR 15-29 mL/min/1.73m^2), and individuals with stage 1, 2, or 3 CKD (eGFR grearter than or equal to 30 mL/min/1.73m^2). Therapy for individuals with stage 4 CKD is a particularly compelling unmet need, as many therapies become problematic (e.g. calcineurin inhibitors will further lower GFR and intensification of renin-angiotensin-aldosterone system inhibitors may lower GFR and raise serum potassium levels). eGFR will be assessed using serum creatinine (Cr) and cystatin C (CystC) using the CKD-EPI Cr/CystC equation for adults.
  7. Subjects must be able to comply with requirements of the protocol, including blood collection, drug administration, and effective communication with study staff.
  8. Heterosexual couples must use at least one effective form of birth control, unless a hysterectomy, tubal ligation, or vasectomy has been performed. These may include the following: barrier methods, oral or an injection (for example, Norplant or Depo-Provera) contraception medication, and intrauterine devices.

     EXCLUSION CRITERIA:

  <!-- -->

  1. Unwilling or unable to provide informed consent.
  2. Subject who requires use of intravenous diuretics to control edema, as this may result in fluid shifts between the intravascular space and the remainder of extracellular fluid volume. Oral diuretics will not be exclusionary, and we reserve the option to use intravenous diuretics during the study if this becomes necessary.
  3. Subject has a psychiatric illness or neurological disease that would interfere with the ability to comply with the requirements of this protocol. This includes, but is not limited to, uncontrolled/untreated psychotic depression, bipolar disorder, schizophrenia, substance abuse or dependence, antisocial personality disorder, panic disorder, or behavioral problems, which interfere with effective communication.

  4 Vulnerable subjects, including those with impaired cognitive function or are incarcerated will be excluded;

  5. Compromised venous access, such that it would interfere with peripheral intravenous access suitable for taking blood samples.

  6. Subject has a severe disease manifestation that would interfere with the ability to comply with the requirements of this protocol.

  7 Subjects with a positive HIV test including antibody or viral load.

  8. Individuals whose blood contains HBV surface antigen or HCV antibody.

  9. Subject has hepatic laboratory parameters (AST, ALT, GGTP) greater than 3 times the upper limit of normal.

  10. Subject is anemic with hematocrit .less than or equal to 30 (for both men and women).

  11. Subject shows evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic (including diabetes mellitus), or gastrointestinal disease, or has a condition that requires immediate surgical intervention.

  12. Subject is pregnant or breastfeeding at any time during the study.

  13. Subject has received treatment with another investigational drug, investigational device, or approved therapy for investigational use less than 60 days prior to ManNAc dosing.

  14. Subject has a hypersensitivity to ManNAc or in the judgment of the investigator, has a condition that places the subject at increased risk for adverse effects.

  15. Subject has been treated with ManNAc, sialic acid, intravenous immunoglobulin (IVIG), and/or other supplements containing sialic acid (e.g., St. John s Wort, sialyllactose) less than 60 days prior to planned ManNAc dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
To assess safety by self-reported symptoms and by standard laboratory testing | in-patient stay by lab results
  Safety by self-reported symptoms and by standard laboratory testing. The effects of reduced eGFR will be assessed. The effect of ManNAc therapy on proteinuria, from the baseline to the end of the extension phase, will be examined on a research basis.

SECONDARY OUTCOMES:
The effects of low serum albumin and reduced eGFR will be assessed. | Baseline to the end of the extension phase
  Subjects are recruited and grouped by eGFR and ManNAc dose. The effects of reduced eGFR on these parameters will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Kopp, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huizing M, Ganguli A, Bolanos J, Leoyklang P, Wilkins KJ, Zeng Y, Figg WD, Rossignol F, Malicdan MCV, Kopp JB, Gahl WA; NIH-ManNAc Study Team. Phase 1 Study of Oral N-Acetylmannosamine in Primary Podocytopathies. Kidney Int Rep. 2025 Dec 31;11(3):103758. doi: 10.1016/j.ekir.2025.103758. eCollection 2026 Mar. PMID 41630898
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-DK-0036.html